CLINICAL TRIAL: NCT06297954
Title: Usefulness of Metoclopramide to Improve Endoscopic Visualization in Upper Gastrointestinal Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Jose Luis Herrera Elizondo, Principal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GA22-00011
Record Dates: First submitted 2024-02-23; First posted 2024-03-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Metoclopramide; Endoscopy; Hematemesis; Melena
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hematemesis; Melena | interventions — Metoclopramide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive metoclopramide 20 mg IV or placebo, this randomization will be performed by means of a computer sequence to receive each of the treatment sequences. The sequence of treatment (metoclopramide) and placebo in which they will be distributed to patients will be determined using randomization software. A folio number will be assigned and depending on the sequence the treatment or placebo will be administered. Subsequently, the upper endoscopy will be performed in the following 120 minutes, and the endoscopic visualization will be evaluated by the physician performing the procedure by means of the modified Avgerinos scale
Who Masked: Participant, Care Provider
Masking Description: As it is double-blind, both physician and patient will not know the treatment they are receiving and it will only be revealed later at the end of the protocol. Following the previous folios, both the treatment and the placebo will be distributed in boxes by default by the research staff, delivering them to the personnel who will apply the drug or placebo, indicating the doses and frequencies of these when administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metoclopramide (Experimental): Patients will be randomized to receive metoclopramide 20 mg IV single dose.
  Interventions: Drug: Metoclopramide
- Placebo (Placebo Comparator): Patients will be randomized to receive placebo 10 ml IV single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide — Patients will receive metoclopramide 20 mg IV in a single dose prior to randomization.
  Arms: Metoclopramide
Drug: Placebo — Patients will receive placebo 10 ml IV in a single dose prior to randomization.
  Arms: Placebo

SUMMARY:
A prospective, randomized, double-blind study will be conducted, including all patients with upper gastrointestinal bleeding, defined as vomiting blood or black bowel movements, within 24 hours prior to admission. Patients will be randomized to receive intravenous metoclopramide 20 mg or placebo, a placebo is a look-alike substance that contains no active drug. Then endoscopy will be performed in the following 120 minutes, evaluating endoscopic visualization with the modified Avgerinos scale.

DETAILED DESCRIPTION:
A prospective, longitudinal, randomized, double-blind study will be carried out in which all patients who come to the University Hospital "Dr. José Eleuterio González" with upper gastrointestinal tract bleeding, defined in our study as hematemesis or melena, including patients with this condition in the 24 hours prior to admission. Patients will be randomized to receive metoclopramide 20 mg IV or placebo, this randomization will be performed by means of a computer sequence to receive each of the treatment sequences. Subsequently, the upper endoscopy will be performed in the following 120 minutes, and the endoscopic visualization will be evaluated by the physician performing the procedure by means of the modified Avgerinos scale; which gives a score of 0-2 according to the percentage of mucosal vision; 0= <25% visible surface, 1= 25%-75% visible surface and 2= >75% visible surface, evaluating fundus, body, antrum and bulb, a score ≥ 6 will be considered a clean stomach and a score ≤ 5 will be considered full stomach. The diagnosis of origin of the upper gastrointestinal tract bleeding will be determined by the physician in charge of performing the endoscopy. All cases will be filmed and another physician will review the cases and validate the Avgerinos score, as well as the final diagnosis reported.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients ≥18 years of age with variceal and non-variceal upper gastrointestinal tract bleeding (hematemesis and/or melena).
* ≤12 hours of bleeding evolution.
* Hemodynamic stability at the time of upper endoscopy.

Exclusion Criteria:

* Patients <18 years old.
* Pregnant patients.
* Metoclopramide allergy.
* Refusal to be part of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
To determine the usefulness of metoclopramide in improving endoscopic visualisation in patients with upper gastrointestinal bleeding. | From admission to discharge for up to 5 days, during this time their clinical condition will be evaluated, through a general physical examination, taking vital signs and questioning them about possible side effects associated with metoclopramide
  Using modified Avgerinos scale; which gives a score of 0-2 according to the percentage of mucosal vision; 0 = <25% visible surface, 1 = 25%-75% visible surface and 2= >75% visible surface, evaluating fundus, body, antrum and bulb, a score ≥ 6 will be considered a clean stomach and a score ≤ 5 will be considered full stomach.

SECONDARY OUTCOMES:
To determine whether the use of metoclopramide avoids repeating the endoscopic procedure. | From admission to discharge for up to 5 days, during this time it will be evaluated the need for new endoscopy in case clinical data of new bleeding from the digestive tract evidenced by melena or hematemesis.
  The need to repeat the endoscopic procedure will be evaluated in case clinical data of new bleeding from the digestive tract, evidenced by melena or hematemesis is found.
To determine whether the use of metoclopramide shortens the length of hospital stay. | From admission to discharge for up to 30 days, during this time their clinical condition will be evaluated, through a general physical examination, taking vital signs and questioning them about possible side effects associated with metoclopramide.
  The days of hospital stay will be counted and comparing both arms.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Herrera Elizondo, Physician, Principal Investigator — Hospital Universitario Dr. José Eleuterio González, UANL
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, UANL, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Estes DJ, Berera S, Deshpande AR, Sussman DA. Re-Visiting Metoclopramide to Optimize Visualization with Gastrointestinal Bleeding - Mobilizing Existing Data. Clin Endosc. 2019 Sep;52(5):516-517. doi: 10.5946/ce.2019.046. Epub 2019 Jul 16. No abstract available. PMID 31309766